CLINICAL TRIAL: NCT07078825
Title: The Effect of Metaverse- and Virtual Reality-Supported Education in the Digital Breastfeeding Museum on Mothers' Breastfeeding Knowledge Level, Self-efficacy, and Success
Brief Title: Metaverse- and VR-Supported Education in the Digital Breastfeeding Museum: Effects on Knowledge, Self-Efficacy, Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Aysenur Akkaya Gul, Instructor, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UU-25-DIGI-BF-MUSE/AAKKAYAGUL
Record Dates: First submitted 2025-07-12; First posted 2025-07-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Metaverse; Virtual Reality; Museum; Breastfeeding Education; Breastfeeding Self-Efficacy
Keywords: Breastfeeding Knowledge Level, Breastfeeding Success

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized controlled trial consisting of two parallel groups: an intervention group receiving Metaverse- and VR-supported education in the digital breastfeeding museum, and a control group receiving standard antenatal class education.
Who Masked: Outcomes Assessor
Masking Description: The statistician performing the data analysis was blinded to the participants' group assignments to prevent bias. No masking was applied; both participants and researchers were aware of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Antenatal Class Education Program Group (No Intervention): No additional intervention was administered to the pregnant women in this group; they only received the routine breastfeeding education provided by the antenatal education program.
- Training Supported by Metaverse and VR in the Digital Breastfeeding Museum Group (Experimental): The pregnant women in this group received training supported by Metaverse and virtual reality (VR) in the digital breastfeeding museum. No additional drugs or medical devices were used throughout the study. The sole intervention consisted of a digital breastfeeding educational program delivered via virtual reality and Metaverse platforms. All content was accessed exclusively through head-mounted displays, without the need for any pharmacological agents or invasive procedures.The environment was explored by participants using virtual reality (VR) headsets (Meta Quest 2).
  Interventions: Other: Training Supported by Metaverse and Virtual Reality (VR) in the Digital Breastfeeding Museum Group

INTERVENTIONS:
Other: Training Supported by Metaverse and Virtual Reality (VR) in the Digital Breastfeeding Museum Group — The pregnant women in this group received training supported by Metaverse and virtual reality (VR) in the digital breastfeeding museum. The training began when pregnant women wore VR headsets (Meta Quest 2) and entered the digital museum using hand controllers. To prevent physical risks like falling or bumping, they navigated the environment safely from where they were seated. Educational content was accessed via personalized avatars. Participants moved between rooms by walking virtually or clicking on circular transition portals. The researcher provided guidance when needed. Video durations varied by topic, totaling around 40 minutes. Mothers could rewatch videos and pause/resume the training on the same day. They engaged with visual, auditory, and written materials, spending approximately one hour in the museum.
  Arms: Training Supported by Metaverse and VR in the Digital Breastfeeding Museum Group

SUMMARY:
This randomized controlled study aimed to evaluate the effect of Metaverse- and virtual reality (VR)-supported education provided in a digital breastfeeding museum on breastfeeding knowledge level, self-efficacy, and breastfeeding success in primiparous pregnant women. The study population consisted of primiparous women who applied for the first time to the antenatal classes of three hospitals in Turkey between July 2023 and April 2024 during their third trimester and had no prior breastfeeding experience. A total of 53 primiparous pregnant women were randomly assigned to the intervention group (n=28) and the control group (n=25). While the intervention group received Metaverse- and VR-supported breastfeeding education in the digital breastfeeding museum, the control group received standard antenatal education provided in routine antenatal classes. Data were collected using a questionnaire assessing participant satisfaction and breastfeeding knowledge, the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), and the LATCH Breastfeeding Assessment Tool. Assessments were performed at three time points: before the intervention, after the intervention, and postpartum.

DETAILED DESCRIPTION:
Breastfeeding is the most ideal way to ensure healthy growth and nutrition for infants. Breast milk is naturally produced to meet the nutritional needs of a newborn. With its unique composition tailored to the specific needs of the developing infant, breast milk is the most appropriate source of nutrition for newborns. Currently low breastfeeding rates are considered a major public health concern. Therefore, promoting breastfeeding is a public health priority. Recognized globally as a fundamental source of nutrition for nearly all infants, breastfeeding gains further importance due to its short- and long-term benefits. Given that breastfeeding benefits not only the baby but also maternal health, providing breastfeeding support to mothers has long been a focus of many national and international health organizations.

In the 21st century, emerging technologies offer alternative educational approaches. These technologies add new dimensions to the learning process and provide more effective educational methods. Virtual reality (VR), with its ability to digitally model the physical world, is one of the technologies used in supplementary education and training. VR refers to computer-generated simulations of real-life environments or scenarios. The Metaverse, on the other hand, is a digital universe where individuals interact through personalized avatars. A review of the literature reveals that there are very few studies using VR technology in breastfeeding education; only two studies have been found to provide such training. No studies were found using a Metaverse-based approach.

This study explores the potential of Metaverse and VR technologies in the field of education and introduces an innovative method for breastfeeding education. Aiming to fill the gap in the literature, a Metaverse- and VR-supported digital breastfeeding education museum was designed as an innovative educational tool for both mothers and educators. The educational content consists of instructional videos, informative written boards, and educational visuals. This material has the potential to offer pregnant women multimodal learning opportunities through visual, auditory, and written channels. Compared to traditional methods, this innovative approach can make education more engaging, increase satisfaction levels, enhance knowledge, improve self-efficacy, and thereby support breastfeeding success.

This study aims to determine the effects of Metaverse- and virtual reality-supported education in a digital breastfeeding museum on mothers' breastfeeding knowledge, self-efficacy, and success. The study was designed as a randomized controlled experimental study. The sample consisted of primiparous pregnant women who applied for the first time to antenatal education programs at three hospitals in Turkey between July 2023 and April 2024, during their third trimester, and had no prior breastfeeding experience. Participants were randomly assigned to groups using a simple randomization method. A total of 53 primiparous pregnant women were randomly assigned to the intervention group (n=28) and control group (n=25). While the intervention group received Metaverse- and VR-supported training in the digital breastfeeding museum, the control group received the routine antenatal education program.

The educational material of the study was the Metaverse- and VR-supported digital breastfeeding museum. A VR web platform (an online virtual reality application enabling interaction through avatars) was used to develop the educational material, allowing users to create 3D virtual environments, provide interactive content, and interact with other users in real time. This platform offered a Metaverse universe that users could explore through their avatars. Through the web platform, a digital museum environment was created, consisting of six different educational rooms: basic principles of breastfeeding, breast milk production and secretion process, breastfeeding positions and considerations during breastfeeding, implementation of breastfeeding and evaluation criteria, milk expression techniques and storage methods, and breastfeeding-related problems. This environment could be explored by participants using VR headsets (Meta Quest 2). The museum content consisted of photo frames, written boards, and instructional videos placed on the walls. The educational application began with mothers wearing the VR headset and using hand controllers to enter the virtual museum. Participants accessed educational content through their personalized avatars. They had the opportunity to engage in multimodal learning through visual, auditory, and written content and spent approximately one hour in the museum.

In addition, the routine education program of the institution continued, and both the intervention and control group participants benefited from this program. No additional intervention was applied to the control group; they only received the standard breastfeeding education provided by the antenatal school. As data collection tools, a questionnaire developed by the researcher based on the literature and two assessment instruments-the Breastfeeding Self-Efficacy Scale-Short Form and the LATCH Breastfeeding Assessment Tool-were used. Prenatal data were collected immediately before and after the training, while postpartum data were collected as soon as possible within the first 24 hours after birth.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous pregnant women who have never given live birth or had any breastfeeding experience and who were attending antenatal classes for the first time during their third trimester,
* Pregnant women who voluntarily agreed to participate in the study,
* Pregnant women aged 18 years or older,
* Pregnant women who are literate in Turkish,
* Mothers who gave birth to newborns with normal gestational age and birth weight.

Exclusion Criteria:

* Pregnant women with physical conditions preventing them from breastfeeding,
* Pregnant women with any condition that would prevent them from completing the questionnaire (e.g., intellectual disability, illiteracy),
* Pregnant women who have difficulty communicating (e.g., with hearing, speech, or visual impairments),
* Pregnant women with any illness that may affect milk secretion or breastfeeding (e.g., cancer, active tuberculosis),
* Pregnant women taking medications that may interfere with breastfeeding,
* Mothers whose newborns have conditions that could interfere with sucking (e.g., cleft lip/palate, being on mechanical ventilation, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Knowledge Score | Immediately before the education, immediately after the education, and within the first 24 hours postpartum
  In order to assess mothers' breastfeeding knowledge levels, a 25-item knowledge questionnaire was developed based on a review of the literature. Each question was scored on a 4-point scale, with the total score ranging from 0 to 100. Participants' responses to the questionnaire were evaluated by assigning points only to correct answers. Incorrect, "I don't know," or unanswered items were not scored. Each participant's total knowledge score was calculated based on the number of correct responses, and the knowledge level was treated as a continuous variable. In this study, no cut-off point was defined to categorize participants as "knowledgeable" or "not knowledgeable"; therefore, knowledge level was interpreted based on the increase in total score.
Breastfeeding Self-Efficacy Scale - Short Form (BSES-SF) Score | Immediately before the education, immediately after the education, and within the first 24 hours postpartum
  The Breastfeeding Self-Efficacy Scale is used to assess how confident mothers feel about their ability to breastfeed. The original scale was developed in 1999. In 2003, the scale was shortened to a 14-item version known as the Breastfeeding Self-Efficacy Scale - Short Form (BSES-SF), which is recommended for use in research and practice. The BSES-SF is a 5-point Likert-type scale, with responses ranging from 1 ("Not at all confident") to 5 ("Always confident"). The minimum possible score is 14, and the maximum is 70. Higher scores indicate higher levels of breastfeeding self-efficacy. The Turkish validity and reliability study of the scale was conducted in 2010. In this study, the Cronbach's alpha coefficient was reported as 0.86.
LATCH Breastfeeding Assessment Tool Score | Within the first 24 hours postpartum
  The LATCH Breastfeeding Assessment Tool is used to evaluate whether breastfeeding mothers are correctly breastfeeding their infants. The acronym LATCH represents five assessment criteria based on the initial letters of the following components:
  * L (Latch on the breast): How well the infant latches onto the breast
  * A (Audible swallowing): Audible swallowing sounds from the infant
  * T (Type of nipple): The type of the mother's nipple
  * C (Comfort breast/nipple): The mother's level of breast/nipple comfort
  * H (Hold): The mother's positioning and ability to hold the baby during breastfeeding
  Each item is scored on a scale from 0 to 2, with a maximum total score of 10. Higher scores indicate greater breastfeeding success. The reliability of the Turkish version of the scale was reported with a Cronbach's alpha coefficient of 0.95.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa, Nilufer, 16059, Bursa, Nilufer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) may be shared upon reasonable request."

REFERENCES:
- [Background] Kilic U, Arar M, Oruc MA. The effect of virtual reality on the breastfeeding process: a randomized controlled study. J Perinatol. 2024 Nov;44(11):1611-1616. doi: 10.1038/s41372-024-02077-0. Epub 2024 Jul 31. PMID 39085438
- See also: Related Info — https://doi.org/10.1038/s41372-024-02077-0
- Available data/document: Publication: 39085438 — https://doi.org/10.1038/s41372-024-02077-0 — This publication provides background data related to the current study's hypothesis and methodology.